CLINICAL TRIAL: NCT00619970
Title: Is Chronic Abdominal Pain in Pediatric Patients Due to Small Intestinal Bacterial Overgrowth?
Acronym: CAP&SIBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Brynie Collins, Assistant Professor of Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCI-06-00146
Record Dates: First submitted 2008-01-25; First posted 2008-02-21 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Chronic Abdominal Pain; Small Intestinal Bacterial Overgrowth
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Control (Active Comparator): Healthy controls
  Interventions: Procedure: Lactulose Breath Test
- Children receiving Rifaximin (Active Comparator): 2/3 Patients with CAP
  Interventions: Drug: xifaxan; Procedure: Lactulose Breath Test
- Children receiving Placebo (Placebo Comparator): 1/3 patients with CAP
  Interventions: Drug: placebo; Procedure: Lactulose Breath Test

INTERVENTIONS:
Procedure: Lactulose Breath Test — Healthy controls will receive one lactulose breath test to assess for SIBO
  Arms: Healthy Control
Drug: xifaxan — xifaxan 550mg TID x10days
  Arms: Children receiving Rifaximin
Drug: placebo — placebo TID x 10days
  Arms: Children receiving Placebo
Procedure: Lactulose Breath Test — Children with CAP will receive one lactulose breath test to assess for SIBO and one after receiving either Rifaximin or Placebo
  Arms: Children receiving Placebo; Children receiving Rifaximin

SUMMARY:
Chronic abdominal pain (CAP) is an extremely pervasive childhood condition and, like IBS in adults, it is one of the functional bowel disorders without a clear framework of understanding or an effective treatment. However, new research suggests that small intestinal bacterial overgrowth (SIBO) may be the unifying pathophysiology that explains the variety of symptoms experienced by patients with IBS. As CAP in children is believed to be a precursor to IBS in adults, we hypothesize that children with this disorder have a significantly greater prevalence of small intestinal bacterial overgrowth (SIBO) than normal, healthy children, and that eradication of bacterial overgrowth with antibiotics will reduce symptoms of chronic abdominal pain in children with this condition. To prove this, we will first aim to determine the prevalence of SIBO in both healthy children and those with CAP. We will do this by performing a lactulose breath hydrogen test, the gold standard for the noninvasive measurement of SIBO, on 40 healthy controls and 80 subjects with CAP. We will then assess whether eradication of SIBO with antibiotics will reduce symptoms of chronic abdominal pain in children with this condition. To do this we will randomize, in a double-blinded fashion, the 80 CAP patients to receive a 10-day course of either the antibiotic Rifaximin or a placebo. After completion of the treatment we will evaluate all these patients for eradication of bacterial overgrowth by repeating a lactulose breath hydrogen test. We will also assess for symptom improvement by re-administering questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 8 and 18
* Subjects must be able to swallow pills
* Healthy Controls must be siblings, other family members or friends of the CAP subjects or children who are undergoing an overnight fast in order to obtain AM labs for another purpose other than this study.
* Female CAP subjects who are sexually active or who may become sexually active during the study will be required to practice an effective method of birth control (e.g., oral contraceptives, contraceptive patch or injection, IUD, double barrier method) before entering into the study.
* All CAP subjects must meet the Rome II Criteria for Functional Bowel Disorders Associated with Abdominal Pain or Discomfort in Children

Exclusion Criteria:

Subjects will be excluded if they:

* have a history of inflammatory bowel diseases, diabetes, cirrhosis or other liver disease, juvenile rheumatoid arthritis, systemic lupus, a history of bowel resection (including gastric, small bowel or colon; gallbladder surgery or appendectomy are NOT exclusion criteria).
* have been treated with antibiotics or probiotics within the past 2 months.
* have a history of TB infection or positive Mantoux test performed at screening
* have a history of allergy to rifampin or rifaximin

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brynie S Collins, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Collins BS, Lin HC. Double-blind, placebo-controlled antibiotic treatment study of small intestinal bacterial overgrowth in children with chronic abdominal pain. J Pediatr Gastroenterol Nutr. 2011 Apr;52(4):382-6. doi: 10.1097/MPG.0b013e3181effa3b. PMID 21240023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control | Children Receiving Rifaximin | Children Receiving Placebo
Started | 40 | 49 | 26
Completed | 40 | 46 | 24
Not Completed | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Children Receiving Rifaximin | Children Receiving Placebo | Total
Number analyzed (Participants) | 40 | 49 | 26 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 49 | 26 | 115
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 37 | 18 | 80
  Male | 15 | 12 | 8 | 35
Region of Enrollment [Number; unit: participants]
  United States | 40 | 49 | 26 | 115

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants at Baseline With SIBO
Time Frame: upon enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Control | Children Receiving Rifaximin | Children Receiving Placebo
Number analyzed (Participants) | 40 | 49 | 26
Participants | 14 | 44 | 24

2. Primary Outcome: Number of Participants With SIBO at Baseline (Week 0) and at 2 Week Post Treatment
Time Frame: baseline (week 0) and at 2 weeks post treatment
Population: 1 patient from the treatment group withdrew from the study. Four additional children, 2 from the treatment group and 2 from the placebo group, did not show up for their follow up breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Children Receiving Rifaximin | Children Receiving Placebo
Number analyzed (Participants) | 49 | 26
Participants
  At baseline | 44 | 24
  2 weeks: number analyzed (Participants) | 46 | 22
  2 weeks | 37 | 19

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Healthy Control | Children Receiving Rifaximin | Children Receiving Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/49 | 0/26
Other Adverse Events (participants affected / at risk) | 0/40 | 0/49 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No